CLINICAL TRIAL: NCT03555487
Title: Clinical Value of 18F -Fluorocholine (18F-FCH) PET in Localizing Parathyroid Lesions: Comparison With 99mTc-sestamibi (MIBI) Scan.
Brief Title: Clinical Value of 18F-FCH PET in Localizing Parathyroid Lesions: Comparison With MIBI Scan.
Acronym: parathyroid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201411046MINB
Record Dates: First submitted 2018-05-20; First posted 2018-06-13 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Parathyroid Diseases
Keywords: Hyperparathyroidism; 18F choline; PET; Tc-99m sestaMIBI; SPECT
MeSH Terms: conditions — Parathyroid Diseases; Hyperparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-choline PET (Experimental): PET/CT
  Interventions: Drug: 18F-choline PET

INTERVENTIONS:
Drug: 18F-choline PET — 5mCi of 18F-FCH will be injected intravenously. PET imaging will be performed on PET/CT scanner. PET/CT from skull base to diaphragm will be started at 50 minutes after the injection.

SUMMARY:
This prospective study aims to

1. compare the detection rates among sonography, MIBI scan and 18F-FCH PET for localization of the parathyroid lesions including adenoma, hyperplasia or carcinoma; evaluate the usefulness of 18F-FCH PET as a second-line tracer in MIBI scan negative patients.

DETAILED DESCRIPTION:
Hyperparathyroidism is a common endocrine disorder. Primary hyperparathyroidism is due to over-secretion of parathyroid hormone and subsequently hypercalcemia, phyophosphatemia and osteoporosis, while secondary hyperparathyroidism is due to physiological secretion of parathyroid hormone by the parathyroid glands in response to hypocalcemia. Surgical approach is the major treatment modality for majority of these patients with hyperparathyroidism. Pre-operative localization of hyperfunctioning glands may lead to minimally invasive surgery. The most commonly used imaging modality for this purpose is 99mTc-sestaMIBI, and supplemented by ultrasonography of the neck. However, the sensitivity and specificity is significantly lower in patients with multiple parathyroid lesions.

Recently, some investigators reported cases of parathyroid adenoma discovered incidentally on choline PET images performed for prostate cancer. 11C or 18F choline is a PET probe used in imaging prostate cancer and hepatocellular carcinoma. As a phospholipid analog, choline is integrated into newly synthesized membranes of proliferating cells by up-regulation of choline kinase. In addition, a previous study showed that the activity of phospholipid/Ca2+-dependent protein kinase was also higher in hyper-functioning parathyroid tissue than in atrophic parathyroid gland. Both mechanisms may be responsible for the uptake of choline tracers in hyperfunctioning parathyroid tissue. Up to now, there are only 3 original reports with limited patients using choline PET in the evaluation of hyperparathyroidism.

This prospective study aims to

1. compare the detection rates among sonography, MIBI scan and 18F-FCH PET for localization of the parathyroid lesions including adenoma, hyperplasia or carcinoma;
2. evaluate the usefulness of 18F-FCH PET as a second-line tracer in MIBI scan negative patients.

ELIGIBILITY:
Inclusion Criteria:

* Parahyperthyroidism (serum iPTH 65 pg / mL; normal range : 12-65), merged with normal or high serum calcium concentration (serum calcium 2.35 mmol / L; normal range: 2.15-2.58) and normal or low serum phosphate concentration (serum phosphorus 3.75 mg / dL; normal range : 2.5-5.0).
* High serum calcium concentration (serum calcium 2.58 mmol/L), but the blood parathyroid hormone concentration in normal range (serum iPTH 12-65pg / mL), hyperthyroidism is suspected.
* MIBI scan has been performed or arranged.
* Age：above 20 years old.

Exclusion Criteria:

* Patient with Familial hypocalciuric hypercalcemia：daily calcium excretion < 100 mg/24h and fractional excretion of calcium < 1%.
* taking or was taking lithium.
* vitamin D deficiency (25-OH vitamin D < 10 ng/mL).
* Patients with pregnancy or recently having a plan for pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
PET imaging | in 3 days
  By visual interpretation if there are focal areas of abnormal 18F-FCH accumulation. The presence, number, size, character, and location of suspected lesions will be filed for each patient in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No